CLINICAL TRIAL: NCT00983632
Title: Selective Vagus Nerve Stimulation in Human
Acronym: VNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Podbregar Matej, Prof., University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VNS
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Arterial Hypertension; Ischemic Heart Disease
Keywords: vagus nerve stimulation; heart rate; systolic arterial pressure
MeSH Terms: conditions — Hypertension; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vagus stimulation (Experimental): electrical vagus stimulation to X.nerve on neck
  Interventions: Procedure: Selective vagus nerve stimulation; Device: selective vagus nerve stimulation

INTERVENTIONS:
Procedure: Selective vagus nerve stimulation — Stimulus will be combination of quasi-trapezoidal cathodic and rectangular anodic current pulses. Precisely, the resulting current, biphasic and charge balanced combination will be composed of a quasi-trapezoidal cathodic phase with a square leading edge with different intensity ic , a plateau tc of 300 μs, and exponentially decaying phase texp of 500 μs, followed by a wide rectangular anodic phase ta of allow current magnitude ia. Anodic phase ia will be one-tenth of the magnitude in the cathodic phase. However, the width of the anodic phase ta will be dependent upon the charge injected in the cathodic phase: the greater the charge, the wider the anodic phase.
  For details see detailed study description
Device: selective vagus nerve stimulation — electrical vagus stimulation

SUMMARY:
The investigators would like to explore possibilities of selective vagus nerve stimulation in human subjects to control heart rate and arterial blood pressure.

DETAILED DESCRIPTION:
Introduction:

The use of nerve stimulation for treating and controlling a variety of medical, psychiatric, and neurological disorders has seen significant growth over the last several decades. In particular, vagal nerve stimulation (VNS) has been the subject of considerable research.

The vagus nerve extensively innervates the thoracic and abdominal viscera (afferent 80% of fibres) and is an important route of information into the central nervous system (efferent 20% of fibres). One of the vagus main functions is to monitor and control the activity of the internal organs and glands such as the heart, lung, stomach, bladder and pancreas.

Activation of the parasympathetic pathway leads to negative chronotropic, negative dromotropic, and negative inotropic changes in the heart. 11 The postganglionic neurons in the vagus nerve project to the sinoatrial (SA) and atrioventricular (AV) nodes, as well as to the atrial and ventricular musculature. In the adult, the right vagus nerve innervates predominantly the SA node, the atrial muscle and, to a much lesser degree, the AV node. On the other hand, the left vagus nerve innervates the SA node and atrial muscle to a lesser degree than it innervates the AV node. However, there can be significant overlap in the anatomical distribution.

Stimulation of the right vagus slows the rate of discharge of the pacemaker cells in the SA node thus slows the SA node rate and thereby reduces the HR. Stimulation of the left vagus nerve produces some slowing of the SA node, prolongation of AV conduction and partial or total AV block. Detailed human data of the vagus nerve stimulation and its effects on heart rate are not available.

The aim of present study is to find clinically acceptable frequency of biphasic VNS, which could allow gradual decrease of heart rate and systemic arterial pressure.

Methods:

Patients undergoing carotid end-arterectomy and coronary bay-pass surgery will be included in the study. Study was approved by The National Medical Ethics Committee, Ministry of Health, Republic of Slovenia (No. 142/02/07, 13 February 2007). Before any trial activity will be performed, the Informed Consent in accordance with the Informed Consent Procedure will be properly obtained.

Design of a Multi-electrode Spiral Cuff:

The self-sizing spiral design was chosen for the cuff. A detailed description of the 39-electrode cuff, having thirteen circumferential groups of three electrodes (GTE 1-13) and fabrication can be found in our previous report.

Anesthesia:

One hour before surgery, patients will be premedicated orally with diazepam 5 mg and pantoprazole 40 mg. For induction into anesthesia short-acting intravenous anaesthetic agent propofol will be used in doses 1 - 2 mg/kg of body weight (BW) administered as a slow bolus doses (20 - 30 s), while remifentanyl (Ultiva, GlaxoSmithKline, GSK Export VB) as a short-acting synthetic μ-opioid agonist will be used in initial loading dose of 1 - 1.5 µg/kg of BW administered in 30 to 60 s period.To facilitate endotracheal intubation a muscle relaxant vecuronium bromide will be administered intravenously.

For maintenance of general anesthesia an inhalation anesthetic isoflurane will be used in inspired concentrations of 1.5 to 3.0 % and analgesia will be assured by a continuous infusion of 0.3 - 0.5 µg/kg/min of remifentanyl. Vecuronium bromide will be administered if muscle relaxation of higher degree was needed of any reason. Low-flow anesthetic technique will be performed by further continuously inhaled fresh gas flow up to 1.5 L/min of oxygen and air mixture to reach 40% of FiO2. Patients will be mechanically ventilated with predetermined tidal volume (VT) (5 - 7 ml/kg of BW), positive end-expiratory pressure (PEEP) between 3 - 5 cm H2O and respiratory rate (RR) between 12 and 15 per minute to maintain ETCO2 between 30 and 35 mm Hg.

During maintenance, an excessive decrease of systemic blood pressure occurred due to depth of anesthesia, was corrected by lightening anaesthesia. To avoid eventual myocardial ischemia, maintenance of normal haemodynamics was strictly controlled.

ECG Recording:

ECG from the first bipolar limb lead (Lead I) will be recorded via self-adhesive, disposable and pre-gelled Ag/AgCl Monitoring Electrode.

Haemodynamic monitoring:

Pressure at airway opening (Pao) will be monitored using a transducer for invasive blood pressure monitoring and attached to a cuffed endotracheal tube. Invasive systemic arterial pressure (SAP) will be measured by the same transducers attached to intra-arterial line placed in left or right radial artery. The central venous catheter for central venous pressure (CVP) and Swan-Ganz catheter (Swan-Ganz CCOmbo Pulmonary Artery Catheter and Vigilance II Monitor, Edwards Inc., USA) for continuous cardiac output and pulmonary artery pressure (PAP) measurements will be inserted after the induction into general anesthesia via right jugular internal vein.

All signals were amplified by a custom designed battery powered bridge amplifier with an adjustable gain. All amplified signals, including amplified ECG, will then be fed to a high-performance data acquisition A/D converter for notebook PC. Data will be stored on a personal computer hard drive for off-line reanalysis. Graphical presentations of results will be performed using the AxoScope 10.2, software developed by Axon Instruments, Inc., 3280 Whipple Road, Union City, CA 94587 USA.

Cuff implantation:

After internal carotid endarterectomy and off-pump coronary artery by-pass surgery cuff around left vagus nerve will be implanted. The vagus nerve passes vertically down the neck within the carotid sheath, lying between the internal jugular vein and internal carotid artery as far as the upper border of the thyroid cartilage, and then between the same vein and the common carotid artery to the root of the neck. The further course of the nerve differs on the two sides of the body.

The vagus nerve will be identified in the carotid sheath in a posterior groove between the carotid artery and the jugular vein. Vessel loops will be used to mobilize the vagus nerve so that about 2.5 to 3 cm will be available for attachment of the spiral cuff. After, the nerve segment will be completely freed from its surrounding tissues and the cuff was then carefully attached to the exposed nerve. Since the need to "seal" the cuff on the nerve with a suture will be unnecessary, the cuff implantation was a relatively simple operation. Namely, the self-fitting nature of the spiral design made it easy to fit snug cuff on a nerve. Furthermore, the spiral cuff design was devised to induce very low pressure when installed on the nerve so that any passively-induced nerve damage will be eliminated. A special care however, will be taken to route the leads to the connector to avoid as much as possible a mechanical tension being transmitted to the cuff. Special care will be taken during surgery also to avoid of causing any mechanical trauma to the recurrent laryngeal nerve.

Vagus nerve stimulation:

Stimulus Stimulus will be combination of quasi-trapezoidal cathodic and rectangular anodic current pulses. Precisely, the resulting current, biphasic and charge balanced combination will be composed of a quasi-trapezoidal cathodic phase with a square leading edge with different intensity ic , a plateau tc of 300 μs, and exponentially decaying phase texp of 500 μs, followed by a wide rectangular anodic phase ta of alow current magnitude ia. Anodic phase ia will be one-tenth of the magnitude in the cathodic phase. However, the width of the anodic phase ta will be dependent upon the charge injected in the cathodic phase: the greater the charge, the wider the anodic phase.

Identification of Particular Nerve Compartments and groups of tree electrodes (GTE) Stimuli with intensity ic of a quasi-trapezoidal cathodic phase of 2 mA with frequency of 20 Hz will be delivered for approximately 10 seconds quasi-bipolarly to all 13 GTEs within the cuff. Stimulation of the separate GTE will be performed 1 minute apart. The GTE that elicited the largest change in heart rate, namely GTE1, will be considered as relevant for further stimulation.

Vagus stimulation with different frequency and increasing current Approximately 10-second long pulse trains with intensities ic of 0.5, 1.0, 1.5, 2.0, 2.5 and 3.0 mA at different frequencies of stimulation (10Hz, 20Hz and 30Hz) will be delivered to aforementioned GTE1 until the absence of cardiac contraction occurred. VNS will be terminated instantly after the absence of cardiac contraction was noticed. The time interval between different two simulations will be at least 2 minute or lasted till heart rate or SAP have not reached basal value before stimulation train. Stimulation will be recorded on the same system as ECG, SAP, PAP, CVP and PAO.

Results:

We expect to find optimal frequency/current relationship of selective VNS which could allow clinical useful manipulation of heart rate and systemic arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing carotid endarterectomy and CABG
* sinus rhythm

Exclusion Criteria:

* acute myocardial infarction
* acute heart failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change of heart rate and blood pressure after vagus nerve stimulation | 1day

CONTACTS AND LOCATIONS:
Overall Officials: Matej Podbregar, PhD MD, Principal Investigator — UMC Ljubljana, Slovenia
Locations (1):
- University medical center, Ljubljana, Slovenija, Slovenia